CLINICAL TRIAL: NCT02204150
Title: Pilot Study for Imaging of the Esophagus Using an OFDI Capsule
Brief Title: Study to Image the Esophagus Using the OFDI Capsule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011P002619; 5R01CA103769-07 (NIH)
Record Dates: First submitted 2014-06-12; First posted 2014-07-30 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Barrett's Esophagus; Eosinophilic Esophagitis
Keywords: Optical Coherence Tomography; Barrett's Esophagus; Esophagus; Imaging
MeSH Terms: conditions — Barrett Esophagus; Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OFDI Capsule Imaging (Experimental): Subject will swallow the OFDI capsule and imaging will be acquired using the OFDI Imaging system.
  Interventions: Device: OFDI Capsule

INTERVENTIONS:
Device: OFDI Capsule — Imaging of the esophagus using the OFDI Capsule and system

SUMMARY:
The main purpose of this research is to test the feasibility and tolerability of the tethered capsule Optical Frequency Domain Imaging (OFDI)

DETAILED DESCRIPTION:
A total of 56 subjects with Barrett's Esophagus, EoE and healthy volunteers will be asked to swallow the OFDI capsule while being unsedated. The capsule is attached to a tether that allows the capsule operator to navigate the capsule as it progresses down the esophagus using natural propulsion called peristalsis as well as to bring it back up to pulled out of the mouth when the procedure is done.

As the capsule progresses down the esophagus, multiple, two dimensional, microscopic cross- sectional images of the esophagus are acquired.

ELIGIBILITY:
Inclusion Criteria:

* A previous diagnosis of Barrett's Esophagus
* OR a previous diagnosis of EoE
* OR a previous diagnosis of Gastroesophageal reflux disease (GERD)
* Subject must be 18 years or older in case of Barrett's and GERD, and over the age of 16 years for EoE
* Subject must be able to give informed consent

Exclusion Criteria:

* Subjects with known esophageal strictures, intestinal strictures or dysphagia
* OR subjects with a history of prior GI surgery or GI Intestinal Crohn's disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD., PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this feasibility study we try to establish the overall number of participants who are able to swallow the capsule and provide us with quality imaging using this new technology. At this point we do no distinguish tolerability separately in each of the three groups and are treating them as one.
Period: Overall Study
Arm/Group | OFDI Capsule Imaging
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OFDI Capsule Imaging
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 38
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of OFDI Imaging in Subjects Swallowing the OFDI Capsule
Description: Number of subjects from whom the quality OFDI imaging was obtained
Time Frame: Images will be acquired during the OFDI imaging session which should take an average of 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | OFDI Capsule Imaging
Number analyzed (Participants) | 56
Participants | 56

ADVERSE EVENTS:
Arm/Group | OFDI Capsule Imaging
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No